CLINICAL TRIAL: NCT06284824
Title: Prospective, Randomized, Single-center Study Comparing the Stryker MAKO™ Robotic-Arm Assisted Total Knee Arthroplasty and the DePuy VELYS™ Robotic-Assisted Solution for Total Knee Arthroplasty.
Brief Title: Comparison of Two Robotic-Assisted Total Knee Arthroplasty Systems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast Orthopedic Specialists (Network)
Collaborators: DePuy Orthopaedics (Industry); Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPS-JMP-2022-040
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Knee Disease
Keywords: robotic assistance; arthroplasty; TKA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MAKO group (Experimental): Patients in this arm will receive the Stryker Triathlon implant and the MAKO robotic arm will be used during surgery.
  Interventions: Device: Stryker Triathlon with MAKO Robotic-Arm
- VELYS group (Experimental): Patients in this arm will receive the DePuy Attune implant and the VELYS robotic arm will be used during surgery.
  Interventions: Device: DePuy Attune with VELYS Robotic-Assistance

INTERVENTIONS:
Device: Stryker Triathlon with MAKO Robotic-Arm — Implant is the Stryker Triathlon total knee arthroplasty and the robotic device is the MAKO robotic-arm
  Arms: MAKO group
Device: DePuy Attune with VELYS Robotic-Assistance — Implant is the DePuy Attune total knee arthroplasty and the robotic device is the VELYS robotic-assistance
  Arms: VELYS group

SUMMARY:
The goal of this prospective study is to compare two different knee replacement robots. This study will look at patient reported outcome measures and data collected during the operation. The main questions this study aims to answer include:

* Will the patient reported outcomes differ between the two groups?
* Will the intraoperative data differ between the two groups? Participants will undergo total knee replacement with one of the two robots, complete standardized surveys, and have x-rays taken.

DETAILED DESCRIPTION:
The purpose of this study is to compare two different total knee arthroplasty (TKA) robotic assisted (RA) devices. This study will compare patient reported outcome measures prior to and after surgery. These surveys will be used determine if there are differences in patient recovery after TKA depending on the robot used. Radiographs will also be taken and used to compare component positioning. Intraoperative data will be collected to compare OR efficiency of the two systems.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a candidate for primary TKA (either Stryker Triathlon with MAKO Robotic-Arm or DePuy Attune with VELYS Robotic-Assistance).
* Individuals who are able to speak, read, and comprehend the Institutional Review Board approved Informed Consent Document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of information to the Sponsor.
* Individuals who are willing and able to complete follow up visits, questionnaires, and radiographic evaluations as specified by the study protocol.
* Individuals who are male or non-pregnant female age 18-80 years at time of device implantation.
* Patient has a diagnosis of primary osteoarthritis or degenerative joint disease of the knee.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) > 40.
* Patient has been diagnosed with osteoporosis or displays poor bone quality per the discretion of the investigator.
* Patient has an active or suspected latent infection in affected knee joint. Patient has neuromuscular or neurosensory deficiency.
* Patient is diagnosed with systemic disease or metabolic disorder (e.g., Lupus, Charcot's. Paget's).
* Subject is a woman who is pregnant or lactating.
* Patient has a contralateral amputation.
* Patient's affected knee has a flexion contracture greater than 15 degrees.
* Patient has history of post operative arthrofibrosis.
* Patient's affected knee has a partial knee arthroplasty.
* Patient has undergone contralateral TKA within the last three months.
* Patient is currently involved in any personal injury litigation, medical-legal, or worker's compensation claims.
* Patient who is bedridden per the discretion of the investigator.
* Patient has a medical condition with less than 2 years of life expectancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
KSS | baseline
  Knee Society Score
KSS | 6 week
  Knee Society Score
KSS | 12 week
  Knee Society Score
KSS | 1 year
  Knee Society Score
KOOS JR | baseline
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement
KOOS JR | 6 week
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement
KOOS JR | 12 week
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement
KOOS JR | 1 year
  Knee injury and Osteoarthritis Outcome Score for Joint Replacement
FJS-12 Knee | 6 week
  Forgotten Joint Score
FJS-12 Knee | 12 week
  Forgotten Joint Score
FJS-12 Knee | 1 year
  Forgotten Joint Score

SECONDARY OUTCOMES:
Operative step time | Intraoperative
  Timing for use of robot during surgery

OTHER OUTCOMES:
Bone resected | Intraoperative
  Amount of bone resected
Costs for surgery | Immediate post operative
  Factors associated with insurance costs for surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Redmond, MD, Principal Investigator — Southeast Orthopedic Specialists

IPD SHARING:
Plan to Share IPD: No